CLINICAL TRIAL: NCT02251080
Title: Attention Deficit/Hyperactivity Disorder (ADHD) Internet Survey Study in a College Student Population
Brief Title: Attention Deficit/Hyperactivity Disorder Internet Survey Study in a College Student Population
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 00026657
Record Dates: First submitted 2014-09-24; First posted 2014-09-26 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2015-12

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: adherence; internet-based
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Internet-based Survey: Assessments completed over the 2-month study will include: disease severity as measured by DSM-V classification and by several validated measures including the ADHD Rating Scale IV with adult prompts, and Clinical Global Impressions, severity and improvement scales; adherence measures (MEMS® and pill counts); validated medication satisfaction measure (the Treatment Satisfaction Questionnaire for Medication); and quality of life measured using the validated WHO Quality of Life Brief measure (WHOQOL-BREF); and responses to a weekly Internet-based questionnaire of adherence and disease severity.
- Standard-of-Care: Assessments completed over the 2-month study will include: disease severity as measured by DSM-V classification and by several validated measures including the ADHD Rating Scale IV with adult prompts, and Clinical Global Impressions, severity and improvement scales; adherence measures (MEMS® and pill counts); validated medication satisfaction measure (the Treatment Satisfaction Questionnaire for Medication); and quality of life measured using the validated WHO Quality of Life Brief measure (WHOQOL-BREF);

SUMMARY:
Attention Deficit/Hyperactivity Disorder (ADHD) is a common condition in young adults. There are many safe oral therapies that require daily use to be effective. Because frequent follow-up visits have been shown to increase adherence to medication, we will determine if adherence to oral therapy for ADHD will improve with an intervention involving weekly internet-based contact without an office visit.

The primary aim is to determine the effectiveness of an Internet-based survey in improving adherence to therapy for ADHD. Subjects in this study will be either receive a weekly Internet-based survey assessing the prescribed medication and their ADHD, or to receive standard-of-care therapy in which they will take their medication. The following hypothesis is to be tested: A weekly Internet survey will promote improved adherence to oral ADHD medications.

DETAILED DESCRIPTION:
This is an investigator-blinded, prospective study of subjects diagnosed with ADHD.Forty-four subjects ages 18 years and older will be enrolled. An Internet-based survey will be piloted to evaluate its effect on adherence to oral ADHD medication. Subjects randomized in a 1:1 ratio to the Internet-survey group will log their impression of the state of their disease on a weekly basis. Subjects in both the intervention and control groups will receive standard-of-care medication, stimulants. Adherence to the medication will be assessed using Medication Event Monitoring System (MEMS®) caps, electronic monitors affixed to the medication containers. Investigators and subjects will be blinded to the adherence data until the final (Month 2) treatment visit.

ELIGIBILITY:
Inclusion Criteria:

* Any male or female 18 years or older of age with a diagnosis of mild to severe ADHD by a psychiatrist at Wake Forest University Student Health Clinic
* Use of the Wake Forest University Student Health Clinic Pharmacy to fill medication for ADHD
* Subject is a good candidate to receive a stimulant for the treatment of their ADHD
* Subject is capable of understanding and willing to provide a signed and dated written voluntary informed consent before any protocol specific procedures are performed
* The subject is able to complete the study and comply with study instructions, including attending all study visits
* Will be filling a prescription for ADHD

Exclusion Criteria:

* Subject is less than 18 years of age
* Inability to complete all study-related visits or inability to complete the Internet survey due to inadequate Internet access
* Patients who are homicidal, suicidal, or psychotic
* Female patients whose medications may be harmful during pregnancy must be on an acceptable form of birth control, otherwise they will not be eligible for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 44 male and female subjects ages 18 and over with ADHD and who are filling the medication at the Wake Forest University Student Health Center pharmacy will be eligible for recruitment. Subjects will be recruited from the Wake Forest University Student Health Center at their clinic visit.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Compared measured adherence of Internet survey group to standard-of-care group | after one month; 2 months of commencing the study
  All subjects will be prescribed the standard-of-care treatment for ADHD, a stimulant. Adherence to standard-of-care medication for ADHD will be objectively measured using a bottle fitted with a Medication Monitoring System (MEMS®) cap and the percentage doses taken will be report as outcome.

SECONDARY OUTCOMES:
Measured adherence by the MEMS® cap in relation to the patient reported adherence via the Internet survey | 2 months
  The Internet survey results of all subjects randomized to receive the Internet survey will be compared to their measured adherence by the MEMS® cap.
Change in disease severity | baseline; month 1, month 2
  Using validated measures the assessments will be done at baseline, month1, and month 2(end of study). Disease severity will be measured by DSM-V classification and by the ADHD Rating Scale IV with adult prompts, and Clinical Global Impressions, severity and improvement scales.

CONTACTS AND LOCATIONS:
Overall Officials: Guy K. Palmes, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States